CLINICAL TRIAL: NCT01649349
Title: The Feasibility Study of Dual-Section Nasogastric Tube in Dysphagia Patients
Brief Title: The Feasibility Study of Dual-Section Nasogastric Tube
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Tsung Ju Wu, M.D., Changhua Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 110807; TW201010751 (Registry Identifier: DUAL-SECTION NASOGASTRIC TUBE)
Record Dates: First submitted 2012-06-29; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Stroke; Mouth Neoplasms
MeSH Terms: conditions — Stroke; Mouth Neoplasms

INTERVENTIONS:
Device: two-piece nasogastric tube — one week period

SUMMARY:
The purpose of this studyis to assess the feasibility and safety of novel designed two-piece nasogastric tube.

ELIGIBILITY:
Inclusion Criteria:

* dysphagia
* mouth neoplasms
* stroke
* already use conventional nasogastric tube for at least 2 weeks

Exclusion Criteria:

* unconsciousness patient
* unstable medical condition with needs of closely medical care
* unable to fill in inform consent
* the fixed length was less than 50 or more than 60 centimeter when using conventional nasogastric tube

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | participants will be followed for the duration of hospital stay, an expected average of 1 weeks
  monitor the adverse events like pressure sore, numbers of self-extubation, dislocation of tube, or other unpredictable events.

SECONDARY OUTCOMES:
satisfaction of Dual-Section Nasogastric Tube | participants will be followed for the duration of hospital stay, an expected average of 1 weeks
  using Likert scale for overall satisfaction